CLINICAL TRIAL: NCT05432505
Title: The Role of Ligamentum Teres Tenodesis in the Management of Developmental Dysplasia of the Hip
Brief Title: Ligamentum Teres Tenodesis in Developmental Dysplasia of the Hip
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Obeid Abd Allah, Principal Investigator, Al-Azhar University
Other Study IDs: LTT
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ligamentum teres tenodesis — Identification of ligamentum teres ligamentum teres tenodesis

SUMMARY:
The treatment of developmental dysplasia of the hip (DDH) remains challenging, yet recent advances have refined our understanding of how best to survey for the condition during infancy, minimize complications during early treatment, and refine the selection of patients who can best benefit from hip preservation surgery. The ideal continued target would be to prevent missed hip dislocations or dysplasia during the infant period, prevent avascular necrosis (AVN) during early treatment, and decrease the incidence of total hip arthroplasty in adulthood related to undertreated DDH, The goal of the treatment is to achieve a concentric reduction of the femoral head into the acetabulum.

DETAILED DESCRIPTION:
it is an operative technique to secure the femoral head after reduction in cases of developmental dysplasia of the hip

Operative technique:

The surgery will be accomplished under a general anesthesia.

An addition to the steps of the open reduction, the following were done:

1. Identification of ligamentum teres
2. ligamentum teres tenodesis

ELIGIBILITY:
Inclusion Criteria:

* Patient with Developmental dysplasia of the hip (DDH) with :

  * Age: from 9 months -5 years old.
  * Virgin DDH.
  * Failed closed reduction in the management of DDH.
  * Failed open reduction through medial approach in the management of DDH

Exclusion Criteria:

* • Paralytic hip dislocation .

  * Post septic hip dislocation.
  * Traumatic hip dislocation .
  * Age : below 9 months or above 5 years.
  * Refusal to participate in this study.

Ages: 9 Months to 60 Months | Sex: All
Age Groups: Child
Study Population: The patients will be examined for:
  1. Length of both lower limbs in relation to each other.
  2. Length of both lower limbs according to patient age.
  3. Presence of hump related to the outer surface of the hip
  4. Presence of pain, abnormal gait, Trendlenburg test Radiographic evaluation (antero posterior and frog pelvis views)
  An addition to the steps of the open reduction, the following were done:
  1. Identification of ligamentum teres
  2. ligamentum teres tenodesis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-21 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
modified HHS | 6 months
  score for function of the hip

REFERENCES:
- [Background] Zhang S, Doudoulakis KJ, Khurwal A, Sarraf KM. Developmental dysplasia of the hip. Br J Hosp Med (Lond). 2020 Jul 2;81(7):1-8. doi: 10.12968/hmed.2020.0223. Epub 2020 Jul 6. PMID 32730146
- [Background] Schaeffer EK, Study Group I, Mulpuri K. Developmental dysplasia of the hip: addressing evidence gaps with a multicentre prospective international study. Med J Aust. 2018 May 7;208(8):359-364. doi: 10.5694/mja18.00154. PMID 29716513